CLINICAL TRIAL: NCT02980718
Title: Does Olfactory Training Improve Olfaction in a Population With Normosmia and How is Their Self Assessment of Sense of Smell?
Brief Title: Does Olfactory Training Improve Olfaction in a Population With Normal Sense of Smell?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/837
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: People With Normal Sense of Smell
Keywords: Olfaction training; Smell
MeSH Terms: conditions — Anosmia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intensive olfactory training (Experimental): 90 participants will undergo intensive olfactory training. They will sniff on four selected odors (10 seconds on each odor bottle in a total of 4 minutes) every morning and evening for 3 months and they will be instructed in the principles of the logbook for olfactory training.
  Interventions: Behavioral: intensive olfactory training
- ordinary olfactory training (Experimental): 90 participants will undergo ordinary olfactory training. They will sniff on four selected odors (10 seconds on each odor bottle in a total of 40 seconds) every morning and evening for 3 months and they will be instructed in the principles of the logbook for olfactory training.
  Interventions: Behavioral: ordinary olfactory training
- controls (No Intervention): 20 participants represent a control group with no olfactory training

INTERVENTIONS:
Behavioral: intensive olfactory training
  Arms: intensive olfactory training
Behavioral: ordinary olfactory training
  Arms: ordinary olfactory training

SUMMARY:
Awareness of the sense of smell in the western population has been low. Most people do not think about the consequences of absence of smell (anosmia). Reduction in sense of smell (hyposmia) can influence everyday life. In situations of stress anosmia can be life threatening for example when there is a fire. Cooks may lose their job. Not being able to enjoy food and drink interferes with quality of life. The causes of olfactory dysfunction (OD) vary. Most often OD is associated with upper respiratory tract infections, disease of the nose and sinuses or head injuries. OD may be congenital, age related or associated with neurological disorders. Hyposmia occurs in up to 85% of cases of Parkinson's and may be the first symptom of both Parkinson's and Alzheimer's disease several years before the mental changes occur.

Knowledge and focus on OD has until recently been low among most physicians and treatment options have often not been available. Different approaches to improve OD have been tried with variable effect depending on the cause of OD. There are studies on corticosteroids, zinc gluconate and vitamin A. In recent years, olfactory training has been launched as a promising treatment option. Most studies with olfactory training are done with patients with OD. A recently published review describes 10 studies with olfactory training among 639 patients and concludes that daily stimulation with odorants (odor concentrate) over a limited period time is a promising treatment. The suggested duration of olfactory training varies from 3 to 14 months. Different intensities of olfactory training were compared in patients with post-viral OD. Olfaction was more improved by the high concentration of odorant than by the low concentration.

A small number of studies have shown that the olfactory nerve to some extent can be trained in persons with normal sense of smell, but we need more experience and structured studies to be able to conclude with greater certainty about the effect of olfactory training in this population.

This study examines whether intensive olfactory training improves the sense of smell more than ordinary olfactory training in subjects with normal olfaction (normosmia) and examines self-evaluation of olfactory function.

DETAILED DESCRIPTION:
Sub-study: Part of the participants (45/200) will be included in a pilot study which will be an analytical observational study to compare olfactory bulb volume measured on MRI three times during a year, while at the same time resting state fMRI will be measured before and after olfactory training. There is not sufficient data in the literature for power calculations and this sub-study is therefore a pilot study.

ELIGIBILITY:
Inclusion Criteria:

* TDI score > 30.5 measured by Sniffin'Sticks

Exclusion Criteria:

* Not able to follow the olfactory training or follow-up (language, practical implementation, mental condition)
* Disease affecting olfaction (sinusitis, pronounced allergies, recent nasal surgery, Alzheimer's, Parkinson, MS, COPD)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
olfaction assessed by TDI-score according to extended Sniffin'Sticks | 4 months (immediately after completion of the training period)
olfaction self-evaluated and reported in a questionnaire | 4 months (immediately after completion of the training period)

SECONDARY OUTCOMES:
olfaction assessed byTDI-score according to extended Sniffin'Sticks | 1 year (6-7 months after completion of the training period)
olfaction self-evaluated and reported in a questionnaire | 1 year (6-7 months after completion of the training period)

CONTACTS AND LOCATIONS:
Overall Officials: Ståle Nordgård, md prof, Study Director — Norwegian University of Science and Technology; Marit Fagerli, md, Study Director — St Olavs Hospital, Klinikk for Øre Nese Hals
Locations (1):
- St Olavs Hospital, Klinikk ØNH, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katotomichelakis M, Balatsouras D, Tripsianis G, Tsaroucha A, Homsioglou E, Danielides V. Normative values of olfactory function testing using the 'sniffin' sticks'. Laryngoscope. 2007 Jan;117(1):114-20. doi: 10.1097/01.mlg.0000246518.79894.7e. PMID 17202939